CLINICAL TRIAL: NCT06874634
Title: The Impact of Albumin Infusion Targets on Mortality in Patients With Abdominal Sepsis
Brief Title: Albumin Infusion Targets on Mortality in Patients With Abdominal Sepsis
Status: Completed | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2023-470
Record Dates: First submitted 2024-03-11; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: 28-day Mortality
Keywords: sepsis, abdominal infection
MeSH Terms: conditions — Sepsis; Intraabdominal Infections | interventions — Serum Albumin, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HA: serum albumin level was above 35g/L after albumin infusion within 72 hours of ICU admission for intra-abdominal sepsis patients
  Interventions: Drug: Human serum albumin injection
- MA: serum albumin level was between 30 and 35g/L after albumin infusion within 72 hours of ICU admission for intra-abdominal sepsis patients.
  Interventions: Drug: Human serum albumin injection
- LA: serum albumin level was less than 30g/L after albumin infusion within 72 hours of ICU admission for intra-abdominal sepsis patients.
  Interventions: Drug: Human serum albumin injection

INTERVENTIONS:
Drug: Human serum albumin injection — Infusion of human albumin injection into patients with abdominal sepsis admitted to the ICU

SUMMARY:
Hypoalbuminemia has been shown to be significantly associated with increased mortality from abdominal sepsis, and early albumin infusion to maintain high serum albumin concentrations may be beneficial for the recovery of patients with abdominal sepsis. However, there have been no reports on whether administering albumin infusion can improve the prognosis, and there is no unified standard for the optimal serum albumin level for exogenous albumin infusion. This study aims to retrospectively collect patients with abdominal sepsis from 2017 to 2022, and divide them into three groups based on their serum albumin levels on the first day of admission to the ICU (D1): high albumin group (HA): albumin level>35g/L, medium albumin group (MA): albumin level between 30-35g/L, low albumin group (LA): albumin level<30g/L, to explore the relationship between different albumin levels and 28 day mortality rate, as well as the corresponding time point fluid balance The effects of vasoactive drug dosage and organ function, mechanical ventilation time, AKI incidence and renal function outcomes, CRRT usage rate, and hospital stay.

DETAILED DESCRIPTION:
Research Background Introduction to Sepsis and Abdominal Sepsis Sepsis is a life-threatening condition characterized by organ dysfunction due to a dysregulated immune response to infection. Abdominal sepsis, originating from intra-abdominal infections, is particularly challenging due to its high morbidity and mortality rates. The mortality rate for abdominal sepsis ranges from 7.6% to 36.0%, and it can reach up to 50% if it progresses to septic shock. The presence of hypoalbuminemia further complicates the clinical course and prognosis of sepsis patients.

Role of Albumin in Sepsis Albumin is a major plasma protein with several critical functions, including maintaining oncotic pressure, transporting various substances, and modulating the immune response. Hypoalbuminemia, defined as serum albumin levels below 30 g/L, is commonly observed in critically ill patients and is associated with increased mortality and morbidity. In sepsis, hypoalbuminemia may result from increased vascular permeability, decreased synthesis, or increased catabolism of albumin. Previous studies have suggested that hypoalbuminemia is an independent risk factor for mortality in abdominal sepsis. However, the specific impact of hypoalbuminemia on mortality in patients with abdominal sepsis remains underexplored.

Objective of the Study Given the high mortality rates associated with abdominal sepsis and the potential impact of hypoalbuminemia on patient outcomes, this study aims to investigate the association between baseline serum albumin levels and 28-day mortality in patients with abdominal sepsis complicated by hypoalbuminemia. The study also explores the specific level of albumin at which mortality is most affected.

Methods Study Design This study was conducted as a retrospective cohort study in a comprehensive ICU with 79 beds at Nanfang Hospital of Southern Medical University. The study was granted exemption from informed consent by the Ethics Committee due to its retrospective nature and was approved under protocol number NFEC-2023-470. The study complied with the Declaration of Helsinki, and all patient data were anonymized to ensure privacy.

Study Population The study included patients aged ≥18 years with abdominal sepsis admitted to the Department of Critical Care Medicine from September 2017 to February 2022. The inclusion criteria were: intra-abdominal infection, sepsis/septic shock, hypoalbuminemia (plasma albumin level <30 g/L upon admission), and infusion of human albumin within 24 hours of ICU admission. Exclusion criteria included: no hospitalization record, readmission to the ICU, ICU stay <24 hours, and conditions requiring albumin therapy (e.g., cirrhosis with ascites, post-liver transplantation, nephrotic syndrome).

Diagnostic Criteria Intra-Abdominal Infections (IAIs): Based on the 2005 Sepsis Consensus, IAIs were diagnosed if clinical manifestations (abdominal pain, systemic inflammatory response) were consistent with IAIs and laboratory tests of intra-abdominal samples met infection criteria. IAIs were confirmed by microbiological culture or surgical findings.

Sepsis-3.0 Criteria: Sepsis was defined as life-threatening organ dysfunction caused by a dysregulated host response to infection. The Sequential Organ Failure Assessment (SOFA) score increase of ≥2 after infection was used as the clinical criterion for sepsis-related organ dysfunction. Septic shock was diagnosed by persistent hypotension requiring vasopressors to maintain a mean arterial pressure (MAP) ≥65 mmHg and serum lactate >2 mmol/L after fluid resuscitation.

Data Collection Demographic and clinical data were collected, including age, gender, BMI, pre-existing conditions, smoking/alcohol history, and etiology. Vital signs, baseline vasopressor doses, laboratory tests (albumin levels at Day 0 and Day 1), fluid balance, albumin infusion doses, and vasopressor doses within 24 hours were recorded. APACHE II and SOFA scores at admission, renal replacement therapy, mechanical ventilation, ICU and hospital length of stay, and 28-day mortality were documented.

Study Endpoints Primary Endpoint: 28-day mortality rate. Secondary Endpoints: Impact of baseline serum albumin on fluid balance, norepinephrine dosage, mechanical ventilation duration, acute kidney injury (AKI) incidence, continuous renal replacement therapy (CRRT) use, and ICU/hospital length of stay.

Statistical Analysis Data were analyzed using SPSS 22.0. Continuous variables were expressed as mean ± SD (normal distribution) or median (IQR25-IQR75) (non-normal distribution), and categorical variables as n (%). Comparisons between survivors and non-survivors were made using independent samples t-tests, Mann-Whitney U tests, and chi-square or Fisher's exact tests. The predictive value of baseline serum albumin for 28-day mortality was assessed using ROC curve analysis, with the optimal cutoff determined by the Youden index. Cox regression analysis identified mortality risk factors, with factors significant at P<0.05 in univariate analysis included in multivariate analysis. Hazard ratios (HR) and 95% confidence intervals (CI) were calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the Intensive Care Department of Southern Hospital of Southern Medical University from September 2017 to June 2022;

Age ≥ 18 years old;

Meeting the diagnostic criteria for abdominal infection;

Patients who meet the diagnostic criteria for sepsis/septic shock;

Complicated with hypoalbuminemia, i.e. plasma albumin<30g/L after admission;

Human serum albumin injection was infused within 24 hours after check-in into the ICU.

Exclusion Criteria:

* Pregnant or lactating women

Patients who have not been able to obtain relevant diagnosis and treatment information after ICU check-in

Patients who repeatedly stay in the ICU

ICU hospitalization time is less than 24 hours

Pathological conditions that require albumin treatment in clinical practice (cirrhosis with ascites, post liver transplantation, intestinal malabsorption syndrome, nephrotic syndrome, burns);

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects of this study were patients with abdominal sepsis who were admitted to the Intensive Care Department of Southern Hospital of Southern Medical University from September 2017 to February 2022
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
28-day mortality | up to 28 days
  Follow-up on the mortality status of patients within 28 days after ICU admission.

SECONDARY OUTCOMES:
Fliuid balance | up to 72 hours after ICU admission
  Record the patient's fluid intake, fluid output at 72 hours after ICU admission，calculate the differences between each pair of times.
norepinephrine equalent doses | up to 72 hours after ICU admission
  doses of vasopressor agents such as norepinephrine, epinephrine, and dopamine at 72 hours after ICU admission.
Indicators of kidney | up to 72 hours after ICU admission
  Record the patient's urine output, serum creatinine, and blood urea nitrogen levels at 72 hours after ICU admission.
Mechanical ventilation time | up to 28 days
  Record the start and end times of mechanical ventilation support, and calculate the difference between the two.
Indicators of liver | up to 72 hours after ICU admission
  Record the levels of ALT (alanine aminotransferase), AST (aspartate aminotransferase), and TBIL (total bilirubin) at 72 hours after ICU admission.
Indicators of lungs | up to 72 hours after ICU admission
  Record the oxygenation index from arterial blood gas analysis within 72 hours after ICU admission.
ICU hospitalization time | up to 1 year
  Record the time of admission to the ICU and the time of discharge from the ICU. Calculate the differences between each pair of times.
total hospitalization time | up to 1 year
  Record the time of hospital admission and the time of hospital discharge. Calculate the differences between each pair of times.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Critical Care Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided